CLINICAL TRIAL: NCT01137708
Title: A Phase 1, Randomized, Open Label, 2-Way Crossover Study To Assess The Effect Of Multiple Dose CP-690,550 On The Pharmacokinetics Of Single Dose Oral Contraceptive Steroids In Healthy Female Subjects
Brief Title: CP-690,550 And Oral Contraception Drug-Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A3921071
Record Dates: First submitted 2010-05-14; First posted 2010-06-04 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: drug interactions; CYP3A; oral contraceptive; anti-rheumatic agents
MeSH Terms: interventions — Ethinyl Estradiol; Levonorgestrel; tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence 1 (Experimental)
  Interventions: Drug: ethinyloestradiol (EE) and levonorgestrel (LN), CP-690,550 + ethinyloestradiol (EE) and levonorgestrel (LN)
- Treatment Sequence 2 (Experimental)
  Interventions: Drug: CP-690,550 + ethinyloestradiol (EE) and levonorgestrel (LN), ethinyloestradiol (EE) and levonorgestrel (LN)

INTERVENTIONS:
Drug: ethinyloestradiol (EE) and levonorgestrel (LN), CP-690,550 + ethinyloestradiol (EE) and levonorgestrel (LN) — Period 1: 30 mcg ethinyloestradiol and 150 mcg levonorgestrel alone Period 2: 30 mcg ethinyloestradiol and 150 mcg levonorgestrel plus 30 mg CP-690,550 after 9 days of CP-690,550 at 30 mg BID
  Arms: Treatment Sequence 1
Drug: CP-690,550 + ethinyloestradiol (EE) and levonorgestrel (LN), ethinyloestradiol (EE) and levonorgestrel (LN) — Period 1: 30 mcg ethinyloestradiol and 150 mcg levonorgestrel plus 30 mg CP-690,550 after 9 days of CP-690,550 at 30 mg BID Period 2: 30 mcg ethinyloestradiol and 150 mcg levonorgestrel alone
  Arms: Treatment Sequence 2

SUMMARY:
This study is designed to assess whether co-administration of CP-690,550 and oral contraceptives will effect the metabolism of the oral contraceptives in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects
* No evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis

Exclusion Criteria:

* Any medical reason which would contraindicate the administration of oral contraceptives
* Clinically significant infections within the past 3 months or history of febrile illness within 5 days
* Positive screening test for Hepatitis B surface antigen, anti Hepatitis C antibody, or human immunodeficiency virus
* Pregnant or nursing women, and women of childbearing potential who are unwilling or unable to use an acceptable method of nonhormonal contraception

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
AUCinf of ethinyloestradiol (EE) and levonorgestrel (LN) | 12 days

SECONDARY OUTCOMES:
AUClast, Cmax, Tmax, and t½ of ethinyloestradiol (EE) and levonorgestrel (LN) | 12 days
Number of adverse events and number of participants with adverse events | 12 days
Changes in complete blood count and serum chemistry profile | 12 days
Changes in vital signs | 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921071&StudyName=CP-690%2C550%20And%20Oral%20Contraception%20Drug-Drug%20Interaction%20Study